CLINICAL TRIAL: NCT00402181
Title: A Phase 2 Multicenter Study of CNTO 328 (Anti IL-6 Monoclonal Antibody) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: An Efficacy and Safety Study of Siltuximab in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012631; C0328T05; 2006-001897-26
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Intravenous; Monoclonal antibody; Siltuximab; Dexamethasone; CNTO 328
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — siltuximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Plan A (Experimental): Siltuximab 6 milligram per kilogram (mg/kg) as intravenous (directly into the vein) infusion once every 2 weeks for 12 cycles and duration of each cycle is 28 days (if participant have complete or partial response) along with dexamethasone (starting from Cycle 2, If participant do not have complete or partial response) 40 mg tablet orally on Day 1 to 4, 9 to 12 and 17 to 20 for maximum 4 cycles after that on Day 1 to 4 up to 12 cycles.
  Interventions: Biological: Siltuximab; Drug: Dexamethasone
- Treatment Plan B (Experimental): Siltuximab 6 mg/kg as intravenous infusion once every 2 weeks along with dexamethasone 40 mg tablet orally on Day 1 to 4, 9 to 12 and 17 to 20 for maximum 4 cycles (duration of each cycle is 28 days) after that on Day 1 to 4 up to 12 cycles.
  Interventions: Biological: Siltuximab; Drug: Dexamethasone

INTERVENTIONS:
Biological: Siltuximab — Siltuximab 6 mg/kg as intravenous infusion once every 2 weeks for 12 cycles and duration of each cycle is 28 days.
  Other Names: CNTO 328
Drug: Dexamethasone — Dexamethasone 40 mg tablet orally on Day 1 to 4, 9 to 12 and 17 to 20 for maximum 4 cycles after that on Day 1 to 4 up to 12 cycles and duration of each cycle is 28 days.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of siltuximab in participants with relapsed (the return of a disease or the signs and symptoms of a disease after a period of improvement.) or refractory (cancer that does not respond to treatment) multiple myeloma (a type of cancer that begins in plasma cells [white blood cells that produce antibodies]).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (when more than one hospital or medical school team work on a medical research study), non-randomized (a clinical trial in which the participants are not assigned by chance to different treatment groups), prospective (study following participants forward in time) safety and efficacy study of siltuximab in participants with relapsed or refractory multiple myeloma. The study consists of 3 Phases: Screening Phase (from first visit until the first dose of study drug), Treatment Phase (from the first dose to the end-of-treatment), and Follow-up Phase (after end-of-treatment until the end of study). The duration of participation in the study for an individual participant will be up to 4 weeks for Screening Phase, approximately 52 weeks for Treatment Phase and until death, lost to follow-up, withdraw of consent or end of study, whichever, comes first for Follow-up Phase. Treatment will be administered on a 28-day cycle. The study is designed with 2 alternative treatment plans. Treatment Plan A: during first 2 cycles siltuximab will be administered alone, dexamethasone may be added to the treatment regimen based on the participant's response to treatment. Treatment Plan B: siltuximab and dexamethasone combination for the duration of the study. The first 14 eligible participants will follow Treatment Plan A and data evaluation will be conducted for participants after 2 cycles of treatment and 2 post baseline disease assessments. If at least one complete response (CR) or partial response (PR) is observed in 14 participants, all subsequent participants will follow Treatment Plan A. However, if no responses (CR or PR) are observed, all subsequent participants will follow Treatment Plan B. The primary efficacy endpoint will be percentage of participants with overall response. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma with relapsed or refractory disease after failing at least 2 prior lines of therapy
* Prior treatment regimen must have included bortezomib (alone or in combination with other agents)
* Measurable secretory disease defined as either serum monoclonal paraprotein (M- protein) greater than or equal to (>=) 1 gram per deciliter (g/dL) or urine monoclonal (light chain) protein (greater than (>) 200 milligram/24 hours)
* Eastern Cooperative Oncology Group (ECOG) performance status score of less than or equal to (<=) 2 - Participants of childbearing potential must use adequate birth control measures, female participants of childbearing potential must have a negative serum pregnancy test at screening

Exclusion Criteria:

* Treatment with systemic cancer therapy (including clarithromycin) or radiotherapy within 30 days before the first dose of study agent - Treatment with nitrosoureas (a group of alkylating agents used as antineoplastic drugs in the chemotherapy) within 42 days before the first dose of study agent
* Major surgery within 30 days before the first dose of study agent or planning to have surgery (except for minor surgical procedures) during the study
* Serious concurrent illness (medical or psychiatric), uncontrolled infection, or significant cardiac disease characterized by significant ischemic coronary disease (an imbalance between myocardial functional requirements and the capacity of the coronary vessels to supply sufficient blood flow) or congestive heart failure (condition in which the heart is unable to pump out sufficient blood to meet the metabolic need of the body) not under medical control, or any uncontrolled medical condition (for example: uncontrolled diabetes), including the presence of clinical laboratory abnormalities, that places the subject at unacceptable risk by participating in the study or confounds the ability to interpret data from the study
* Known to be seropositive (giving a positive result in a test of blood serum) for Human Immunodeficiency Virus (HIV), or active hepatitis A, B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Overall Response | Baseline up to end of study (Day 807)
  The overall response is defined as percentage of participants having confirmed Complete Response (CR) and Partial Response (PR) by using the European Group for Blood and Marrow Transplantation (EBMT) criteria. CR is absence of the original monoclonal protein (M-protein) in serum and urine maintained for a minimum of 6 weeks, and disappearance of soft tissue plasmacytomas. PR is greater than or equal to (>=) 50 percent reduction in the level of the serum M-protein maintained for a minimum of 6 weeks and >= 50 percent reduction in the size of soft tissue plasmacytomas.

SECONDARY OUTCOMES:
Time to Progression (TTP) | Baseline up to end of study (Day 807)
  The TTP is defined as the time interval in days between the date of first administration of study treatment (as monotherapy or as combination therapy) to the date of first documented evidence of confirmed progressive disease (including relapse from CR). CR is absence of the original M-protein in serum and urine maintained for a minimum of 6 weeks, and disappearance of soft tissue plasmacytomas.
Duration of Response | Baseline up to end of study (Day 807)
  The duration of response is defined as the time from initial documented response (Complete Response [CR] or Partial Response [PR]), to the first documented sign of progression. CR is absence of the original M-protein in serum and urine maintained for a minimum of 6 weeks, and disappearance of soft tissue plasmacytomas. PR is >= 50% reduction in the level of the serum M-protein maintained for a minimum of 6 weeks and >= 50% reduction in the size of soft tissue plasmacytomas.
Number of Participants With Immune Response | Day 1 (Cycle 1 [pre-dose]), treatment discontinuation, and every 3 months after the last dose (up to 3 times)
  Immune response is defined as antibody (type of protein that helps to protect the body against foreign matter, such as bacteria and viruses) response to siltuximab.
Percent Change From Baseline in C-Reactive Protein (CRP) Level | Before siltuximab administration in Cycles 1, 2, and 3 on Days 1 and 15; thereafter, on Day 1 of each cycle up to12 cycles
  Percentage change in CRP is equal to CRP at time of measurement minus CRP at baseline divided by CRP at baseline multiplied by 100.
Percent Change From Baseline in C-telopeptide (CTx) Level | Before siltuximab administration on Day 1 of cycles 1, 2, and 3
  Percentage change in CTx is equal to CTx at time of measurement minus CTx at baseline divided by CTx at baseline multiplied by 100.
Percent Change From Baseline in N-telopeptide (NTx) Level | Before siltuximab administration on Day 1 of cycles 1, 2, and 3
  Percentage change in NTx is equal to NTx at time of measurement minus NTx at baseline divided by NTx at baseline multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (13):
- United States (9):
  - Duarte, California
  - Norwalk, Connecticut
  - Indianapolis, Indiana
  - Rochester, Minnesota
  - New York, New York
  - Chapel Hill, North Carolina
  - Pittsburgh, Pennsylvania
  - North Charleston, South Carolina
  - Houston, Texas
- Netherlands (4):
  - Amsterdam
  - Leiden
  - Rotterdam
  - The Hague

REFERENCES:
- See also: A Phase 2 Multicenter Study of CNTO 328 (Anti IL-6 Monoclonal Antibody) in Subjects With Relapsed or Refractory Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=175&filename=CR012631_CSR.pdf